CLINICAL TRIAL: NCT03881098
Title: The Lung PCA: A Multi-Dimensional Atlas of Pulmonary Premalignancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 19-0400.cc
Record Dates: First submitted 2019-03-07; First posted 2019-03-19 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
Keywords: Bronchoscopy; Squamous Cell Carcinoma; Pre-Malignant Lesions; Smoking; Multi-site
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Squamous Cell; Smoking | interventions — Bronchoscopy; Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Squamous Cell Carcinoma Pre-Malignant Lesions (Other): The prospective SCC-PML cohort is envisioned to provide a well-matched group of high-risk subjects that will provide clinically comparable subjects with lesional sites representing progressive and non-progressive disease.
  Interventions: Procedure: Bronchoscopies; Procedure: Sputum Sample; Procedure: Venipuncture

INTERVENTIONS:
Procedure: Bronchoscopies — Bronchoscopy: Your nose, throat, vocal cords and windpipe are sprayed with Lidocaine (numbing medicine) to help keep you from coughing and to numb your airways. A tube with either a white light or the fluorescent light (bronchoscopy) is put down through your nose or mouth into your throat. Your nose, throat, vocal cords and lungs will be checked for any unusual areas while the tube goes down. You might have medicine sprayed into your mouth. You may be given a shot into your vein or muscle to help you be more comfortable.
  Endobronchial Biopsy: Very tiny pieces of lung tissue (about the size of the head of a pin) will be taken from the lining of your lungs using forceps and a small brush. These tissues will be taken to a laboratory and tested.
Procedure: Sputum Sample — Subjects will be asked to perform the early morning spontaneous cough technique over a six-day period to provide for pre-screening evaluations. If moderate atypia is detected in a pre-screening specimen, additional sputum samples will be collected prior to each subsequent bronchoscopy. If this cannot be performed prior to bronchoscopy with adequate results, the sputum collection may be done after bronchoscopy. The sputum will be collected in containers containing Saccomanno's fixative.
Procedure: Venipuncture — Thirty milliliters of blood will be withdrawn from each subject, and the blood will be sent to the biorepository for analysis and storage.

SUMMARY:
This protocol pertains specifically to the prospective lung squamous cell carcinoma pre-malignant lesion (PML) cohort that will form a primary study group for the Lung Pre-Cancer Atlas.

DETAILED DESCRIPTION:
Via pre-screening, subjects at high risk for the development of lung squamous cell carcinoma (SCC) will be identified and enrolled to undergo serial bronchoscopies at 12 month intervals over a 2-3 year period. A variety of specimen types will be collected to support analyses of the genomic and microenvironmental features of these PMLs.

ELIGIBILITY:
Inclusion Criteria

Prerequisites for Inclusion in Either Study Group:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged > 18 years.

Pre-Screening Inclusion Criteria:

Patients that have consented to the pre-screening with any of the clinical histories described below, will be asked to provide a screening sputum sample and undergo a bronchoscopy. The bronchoscopy is contingent on the identification of moderate or worse bronchial epithelial atypia by sputum cytology. Those patients with moderate or worse atypia on sputum cytology will be offered bronchoscopic examination and tissue sampling. If findings from the bronchoscopy meet Main Study Group inclusion criteria, the patients will be offered a chance to enroll in the main study. The following criteria will be used to identify potential pre-screening enrollees:

1. A current or ex-smoker with a > 20 pack-year history of smoking.
2. History of non-small cell lung cancer (stage I, II, or IIIA) with> 10 pack-year history of smoking and no evidence of active disease at least 1 year after definitive treatment.
3. History of head and neck cancer (stage I, II, III, or IVA) with > 10 pack-year history of smoking and no evidence of active disease at least 1 year after definitive treatment.

Main Study Group Inclusion Criteria:

Enrollment in the main study group can occur via two routes. If inclusion criteria described below are already present from results of a prior bronchoscopy the patient may be enrolled directly. The second route will involve evaluation of results obtained in the pre-screening arm. When a prescreening bronchoscopy shows biopsy histologic findings that meet the pre-requisites shown below, the patient will be offered enrollment in the Main Study Group where they will be offered three more bronchoscopic examinations including the baseline bronchoscopy and those performed at one and two years after the baseline bronchoscopy. Note: the pre-screening bronchoscopy cannot represent the main study group baseline bronchoscopy as costs associated with specialized specimen collection in the main study group (single cell processing, etc.) cannot be covered in the pre-screening bronchoscopy. The qualifying additional pre-requisites for enrollment in the Main Study Group are:

1. Participants must be able and willing to undergo a total of at least three bronchoscopies.
2. Prior results from bronchoscopic analyses (via previous results or from pre-screening cohort bronchoscopies) must meet either of the following criteria to qualify patients as potential Main Study Group enrollees:

   * Pre-existing bronchoscopic documentation of persistence of or progression to high grade dysplasia at two or more airway sites.
   * Endobronchial dysplasia (squamous metaplasia/mild dysplasia, score > 3) at > 3 airway sites.
   * High grade bronchial dysplasia (moderate dysplasia or worse, score > 5)

Exclusion Criteria

Patients will not eligible if any one of the following conditions are present:

1. Clinically apparent bleeding diathesis.
2. Cardiac dysrhythmia that is potentially life threatening, such as ventricular tachycardia, multifocal premature ventricular contractions or supraventricular tachycardias with a rapid ventricular response. Well-controlled atrial fibrillation or rare (< 2/minute) premature ventricular contractions are not exclusionary.
3. Hypoxemia (less than 90% saturation with supplemental oxygen) prior to bronchoscopy.
4. Evidence of clinically active coronary artery disease, including myocardial infarction within 6 weeks, anginal chest pain, or poorly controlled congestive heart failure, or any other serious medical condition which would preclude a patient from undergoing a bronchoscopy.
5. Acute bronchitis or pneumonia within 8 weeks, except if these are considered clinically to be possibly a result of lung cancer.
6. Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-12-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Determine Genomic Features of Pre-Malignant Lesions (PML) via Bronchoscopic Biopsy | Start of study to post baseline bronchoscopy, up to two years
  Prospective data collection of histologic specimens for the purposes of reducing lung cancer mortalities.
Determine Microenvironmental Features of Lung Pre-Malignant Lesions (PML) via Bronchoscopic Biopsy | Start of study to post baseline bronchoscopy, up to two years
  Prospective data collection of histologic specimens for the purposes of reducing lung cancer mortalities.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Keith, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Rocky Mountain Regional VAMC, Aurora, Colorado
  - UCHealth - Metro, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No